CLINICAL TRIAL: NCT01696084
Title: Phase III, Multicenter, Randomized, Trial of CPX-351 (Cytarabine:Daunorubicin) Liposome Injection Versus Cytarabine and Daunorubicin in Patients 60-75 Years of Age With Untreated High Risk (Secondary) AML
Brief Title: Phase III Study of CPX-351 Versus 7+3 in Patients 60-75 Years Old With Untreated High Risk (Secondary) Acute Myeloid Leukemia
Acronym: 301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLTR0310-301
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: High Risk Acute Myeloid Leukemia
Keywords: AML; Acute Myeloid Leukemia; high risk AML; secondary AML; AML in elderly
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (CPX-351) (Experimental): Subjects are eligible to receive up to 2 inductions and up to 2 consolidations with CPX-351. The number of inductions and consolidations a subject received depended on response.
  Interventions: Drug: CPX-351
- Arm B (7+3) (Active Comparator): Subjects are eligible to receive up to 2 inductions and up to 2 consolidations with cytarabine and daunorubicin given as a 7 + 3, or 5 days of continuous infusion of cytarabine and 2 days of daunorubicin (5+2, second induction, consolidation courses) therapy. The number of inductions and consolidations a subject received depended on response.
  Interventions: Drug: 7+3 (cytarabine and daunorubicin)

INTERVENTIONS:
Drug: CPX-351 — First induction: 100 units/m2 by 90-minute IV infusion on Days 1, 3, 5. Second induction: 100 units/m2 by 90-minute IV infusion on Days 1 and 3. Consolidation therapy: 65 units/m2 by 90-minute IV infusion on Days 1 and 3.
  Arms: Arm A (CPX-351)
Drug: 7+3 (cytarabine and daunorubicin) — First induction: 7+3 was administered as: cytarabine at a dose of 100 mg/m2/day on Days 1 through 7 by continuous infusion, and daunorubicin at a dose of 60 mg/m2/day on Days 1, 2, and 3.
  Second induction: 5+2 was administered as: cytarabine at a dose of 100 mg/m2/day on Days 1 through 5 by continuous infusion and daunorubicin at a dose of 60 mg/m2/day on Days 1 and 2.
  Consolidation therapy: 5+2 was administered as: cytarabine at a dose of 100 mg/m2/day on Days 1 through 5 by continuous infusion, and daunorubicin at a dose of 60 mg/m2/day on Days 1 and 2.
  Other Names: cytarabine and daunorubicin
  Arms: Arm B (7+3)

SUMMARY:
To confirm the efficacy of CPX-351 compared to 7+3 as first line therapy in elderly patients (60-75 yrs) with high risk (secondary) Acute Myeloid Leukemia. The primary efficacy endpoint will be overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily give informed consent
* Age 60-75 years at the time of diagnosis of AML
* Pathological diagnosis of AML according to WHO criteria (with at least 20% blasts in the peripheral blood or bone marrow)
* Confirmation of:

  * Therapy related AML: t-AML must have a documented history of prior cytotoxic therapy or ionizing radiotherapy for an unrelated disease
  * AML with a history of myelodysplasia: MDSAML must have bone marrow documentation of prior MDS
  * AML with a history of CMMoL: CMMoLAML must have bone marrow documentation of prior CMMoL
  * De novo AML with karyotypic abnormalities characteristic of MDS: de novoAML must have cytogenetics with abnormalities per WHO.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Able to adhere to the study visit schedule and other protocol requirements
* Laboratory values fulfilling the following:

  * Serum creatinine < 2.0 mg/dL
  * Serum total bilirubin < 2.0 mg/dL, patients with Gilbert's Syndrome should contact the medical monitor
  * Serum alanine aminotransferase or aspartate aminotransferase < 3 times the ULN Note: If elevated liver enzymes, above the ULN, are related to disease; contact medical monitor to discuss.
* Cardiac ejection fraction ≥ 50% by echocardiography or MUGA
* Patients with second malignancies in remission may be eligible if there is clinical evidence of disease stability for a period of greater than 6 months off cytotoxic chemotherapy, documented by imaging, tumor marker studies, etc., at screening. Patients maintained on long-term non-chemotherapy treatment, e.g., hormonal therapy, are eligible.

Exclusion Criteria:

* Except for CMMoL, patients with history of myeloproliferative neoplasms (MPN) (defined as a history of essential thrombocytosis or polycythemia vera, or idiopathic myelofibrosis prior to the diagnosis of AML) or combined MDS/MPN are not eligible.
* Acute promyelocytic leukemia [t(15;17)] or favorable cytogenetics, including t(8;21) or inv16 if known at the time of randomization.
* Clinical evidence of active CNS leukemia
* Patients with active (uncontrolled, metastatic) second malignancies are excluded.
* Prior treatment intended for induction therapy of AML; only hydroxyurea is permitted for control of blood counts. For example, a patient with MDS that changes HMA dose and schedule after the diagnosis of AML is excluded. AML-type therapy, such as cytarabine alone (>1g/m2/day) or cytarabine plus an anthracycline as well as prior HSCT are also excluded.
* Administration of any therapy for MDS (conventional or investigational) must be completed by 2 weeks prior to of the first dose of study drug; in the event of rapidly proliferative disease use of hydroxyurea is permitted until 24 hours before the start of study treatment. Toxicities associated with prior MDS therapy must have recovered to grade 1 or less prior to start of treatment.
* Any major surgery or radiation therapy within four weeks.
* Patients with prior cumulative anthracycline exposure of greater than 368 mg/m2 daunorubicin (or equivalent).
* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent obtaining informed consent
* Patients with myocardial impairment of any cause (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (Class III or IV staging)
* Active or uncontrolled infection. Patients with an infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for ≥72 hrs.
* Current evidence of invasive fungal infection (blood or tissue culture); patients with recent fungal infection must have a subsequent negative cultures to be eligible; known HIV (new testing not required) or evidence of active hepatitis B or C infection (with rising transaminase values)
* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or other copper-metabolism disorder

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2012-12-13 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - University of CA San Diego, San Diego, California
  - Stanford University, Stanford, California
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - North Shore LIJ Health System, Long Island City, New York
  - Columbia University, New York, New York
  - Cornell U, Weill Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Services, Winston-Salem, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Baylor Research Insitute, Dallas, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Cancer Center, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec

REFERENCES:
- [Derived] Shimony S, Murdock HM, Keating JH, Tsai HK, Sasi A, Gibson CJ, Faderl S, Wagner A, Dronamraju N, Lin TL, Prebet T, Cortes JE, Uy GL, Lancet JE, Reilly CR, Neuberg DS, Stone RM, Lindsley RC. CPX-351 Selectively Benefits Patients with AML and Myelodysplasia-Related Mutations in the Pivotal Randomized Trial. Blood Adv. 2026 Feb 2:bloodadvances.2025019378. doi: 10.1182/bloodadvances.2025019378. Online ahead of print. PMID 41628350
- [Derived] Cortes JE, Lin TL, Asubonteng K, Faderl S, Lancet JE, Prebet T. Efficacy and safety of CPX-351 versus 7 + 3 chemotherapy by European LeukemiaNet 2017 risk subgroups in older adults with newly diagnosed, high-risk/secondary AML: post hoc analysis of a randomized, phase 3 trial. J Hematol Oncol. 2022 Oct 26;15(1):155. doi: 10.1186/s13045-022-01361-w. PMID 36289532
- [Derived] Cortes JE, Lin TL, Uy GL, Ryan RJ, Faderl S, Lancet JE. Quality-adjusted Time Without Symptoms of disease or Toxicity (Q-TWiST) analysis of CPX-351 versus 7 + 3 in older adults with newly diagnosed high-risk/secondary AML. J Hematol Oncol. 2021 Jul 13;14(1):110. doi: 10.1186/s13045-021-01119-w. PMID 34256819
- [Derived] Lancet JE, Uy GL, Newell LF, Lin TL, Ritchie EK, Stuart RK, Strickland SA, Hogge D, Solomon SR, Bixby DL, Kolitz JE, Schiller GJ, Wieduwilt MJ, Ryan DH, Faderl S, Cortes JE. CPX-351 versus 7+3 cytarabine and daunorubicin chemotherapy in older adults with newly diagnosed high-risk or secondary acute myeloid leukaemia: 5-year results of a randomised, open-label, multicentre, phase 3 trial. Lancet Haematol. 2021 Jul;8(7):e481-e491. doi: 10.1016/S2352-3026(21)00134-4. PMID 34171279
- [Derived] Lin TL, Rizzieri DA, Ryan DH, Schiller GJ, Kolitz JE, Uy GL, Hogge DE, Solomon SR, Wieduwilt MJ, Ryan RJ, Faderl S, Cortes JE, Lancet JE. Older adults with newly diagnosed high-risk/secondary AML who achieved remission with CPX-351: phase 3 post hoc analyses. Blood Adv. 2021 Mar 23;5(6):1719-1728. doi: 10.1182/bloodadvances.2020003510. PMID 33724305
- [Derived] Kolitz JE, Strickland SA, Cortes JE, Hogge D, Lancet JE, Goldberg SL, Villa KF, Ryan RJ, Chiarella M, Louie AC, Ritchie EK, Stuart RK. Consolidation outcomes in CPX-351 versus cytarabine/daunorubicin-treated older patients with high-risk/secondary acute myeloid leukemia. Leuk Lymphoma. 2020 Mar;61(3):631-640. doi: 10.1080/10428194.2019.1688320. Epub 2019 Nov 25. PMID 31760835
- [Derived] Lancet JE, Uy GL, Cortes JE, Newell LF, Lin TL, Ritchie EK, Stuart RK, Strickland SA, Hogge D, Solomon SR, Stone RM, Bixby DL, Kolitz JE, Schiller GJ, Wieduwilt MJ, Ryan DH, Hoering A, Banerjee K, Chiarella M, Louie AC, Medeiros BC. CPX-351 (cytarabine and daunorubicin) Liposome for Injection Versus Conventional Cytarabine Plus Daunorubicin in Older Patients With Newly Diagnosed Secondary Acute Myeloid Leukemia. J Clin Oncol. 2018 Sep 10;36(26):2684-2692. doi: 10.1200/JCO.2017.77.6112. Epub 2018 Jul 19. PMID 30024784
- [Derived] Stein EM, Tallman MS. Emerging therapeutic drugs for AML. Blood. 2016 Jan 7;127(1):71-8. doi: 10.1182/blood-2015-07-604538. Epub 2015 Dec 10. PMID 26660428

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (CPX-351) | Arm B (7+3)
Started | 153 | 156
Completed | 22 | 10
Not Completed | 131 | 146

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (CPX-351) | Arm B (7+3) | Total
Number analyzed (Participants) | 153 | 156 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (4.19) | 67.7 (4.1) | 67.7 (4.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 60 | 119
  Male | 94 | 96 | 190
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 128 | 139 | 267
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was measured from the date of randomization to death from any cause, subjects not known to have died by the last follow-up were censored on the date they were last known to be alive.
Time Frame: From the date of randomization to death from any cause
Population: Intent-to-Treat (ITT) Population: All participants randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (CPX-351) | Arm B (7+3)
Number analyzed (Participants) | 153 | 156
months | 9.56 [6.60 to 11.86] | 5.95 [4.99 to 7.75]

2. Secondary Outcome: Proportion of Subjects With a Response
Description: Complete Remission (CR)
Time Frame: Post Induction
Population: Intent-to-Treat (ITT) Population: All participants randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (CPX-351) | Arm B (7+3)
Number analyzed (Participants) | 153 | 156
Participants | 57 | 40

3. Secondary Outcome: Event-free Survival
Description: All randomized subjects were assessed for event-free survival (EFS). EFS was defined as the time from study randomization to the date of induction treatment failure (persistent disease), relapse from CR or CRi or death from any cause, whichever came first. Subjects alive and not known to have any of these events were censored on thee date they were last examined on study.
Time Frame: From the date of randomization to the date that persistent disease was documented or the date of relapse after CR or death, whichever came first
Population: Intent-to-Treat (ITT) Population: All participants randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (CPX-351) | Arm B (7+3)
Number analyzed (Participants) | 153 | 156
months | 2.53 [2.07 to 4.99] | 1.31 [1.08 to 1.64]

4. Secondary Outcome: Remission Duration
Description: Only subjects achieving CR or CRi were assessed for remission duration.
Time Frame: From the date of achievement of a remission until the date of relapse or death from any cause
Population: Intent-to-Treat (ITT) Population: All participants randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (CPX-351) | Arm B (7+3)
Number analyzed (Participants) | 153 | 156
months | 6.93 [4.60 to 9.23] | 6.11 [3.45 to 8.71]

5. Secondary Outcome: Rate of Achieving Morphologic Leukemia-free State
Description: All randomized subjects with at least 1 evaluable postrandomization bone marrow assessment performed on or after Day 14 after the last induction were assessed for MLFS.
Time Frame: Day 14
Population: Intent-to-Treat (ITT) Population: All participants randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (CPX-351) | Arm B (7+3)
Number analyzed (Participants) | 126 | 119
Participants | 87 | 66

6. Secondary Outcome: Proportion of Subjects Receiving a Stem Cell Transplant
Description: The number and percentage of subjects transferred for HSCT after induction treatment was recorded.
Time Frame: Post Induction
Population: Intent-to-Treat (ITT) Population: All participants randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (CPX-351) | Arm B (7+3)
Number analyzed (Participants) | 153 | 156
Participants | 52 | 39

ADVERSE EVENTS:
Time Frame: Adverse events (AE) recorded from the start of the infusion on Day 1 to the last day of the treatment period. SAE recorded from the start of the infusion on Day 1 to 30 days after completion of the treatment period.
Description: Safety Population: All randomized participants who received at least one dose of study treatment.
Arm/Group | Arm A (CPX-351) | Arm B (7+3)
All-Cause Mortality (participants affected / at risk) | 1/153 | 0/151
Serious Adverse Events (participants affected / at risk) | 90/153 | 65/151
Other Adverse Events (participants affected / at risk) | 152/153 | 151/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (CPX-351) (N=153) | Arm B (7+3) (N=151)
Febrile Neutropenia (Blood and lymphatic system disorders) | 12 | 8
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 2
Cardiac Failure (Cardiac disorders) | 2 | 2
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 4
Myocardial Infarction (Cardiac disorders) | 3 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Cardiotoxicity (Cardiac disorders) | 0 | 1
Cytotoxic Cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Euthyroid Sick Syndrome (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Conjunctival Haemorrhage (Eye disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Small Intestinal Disorders (Gastrointestinal disorders) | 1 | 1
Chron's Disease (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gingival Bleeding (Gastrointestinal disorders) | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Disease Progression (General disorders) | 6 | 6
Multi-Organ Failure (General disorders) | 2 | 4
Chest Pain (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chest Discomfort (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 2 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Alloimmunisation (Immune system disorders) | 1 | 0
Sepsis (Infections and infestations) | 12 | 5
Pneumonia (Infections and infestations) | 10 | 6
Bacteraemia (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 3 | 1
Septic Shock (Infections and infestations) | 2 | 2
Enterococcal Bacteraemia (Infections and infestations) | 1 | 2
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 2
Lung Infection (Infections and infestations) | 0 | 2
Pneumonia Bacterial (Infections and infestations) | 1 | 1
Bacteroides Bacteraemia (Infections and infestations) | 1 | 0
Bronchopulmonary Aspergillosis (Infections and infestations) | 1 | 0
Central Nervous System Infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Enterobacter Bacteraemia (Infections and infestations) | 1 | 0
Escherichia Bacteraemia (Infections and infestations) | 0 | 1
Escherichia Sepsis (Infections and infestations) | 0 | 1
Klebsiella Bacteraemia (Infections and infestations) | 0 | 1
Klebsiella Sepsis (Infections and infestations) | 0 | 1
Mycotic Aneurysm (Infections and infestations) | 1 | 0
Neutropenic Infection (Infections and infestations) | 1 | 0
Pneumonia Fungal (Infections and infestations) | 0 | 1
Pneumonia Pseudomonas Aeruginosa (Infections and infestations) | 0 | 1
Pseudomonal Bacteraemia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Sinusitis Fungal (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1
Streptococcal Sepsis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Transfusion Reaction (Injury, poisoning and procedural complications) | 2 | 0
Brain Herniation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Transfusion-Related Acute Lung Injury (Injury, poisoning and procedural complications) | 1 | 0
Ejection Fraction Decreased (Investigations) | 9 | 9
Enterococcus Test Positive (Investigations) | 1 | 0
Fungal Test Positive (Investigations) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0
Klebsiella Test Positive (Investigations) | 0 | 1
Pseudomonas Test Positive (Investigations) | 1 | 0
Staphylococcus Test Positive (Investigations) | 1 | 0
Stenotrophomonas Test Positive (Investigations) | 1 | 0
Streptococcus Test Positive (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Lactic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Acute Myeloid Leukaemia Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 4 | 0
Central Nervous System Haemorrhage (Nervous system disorders) | 3 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 2
Haemorrhage Intracranial (Nervous system disorders) | 1 | 1
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 2 | 0
Delirium (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 2 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (CPX-351) (N=153) | Arm B (7+3) (N=151)
Febrile Neutropenia (Blood and lymphatic system disorders) | 104 | 105
Atrial Fibrillation (Cardiac disorders) | 8 | 15
Conjunctival Haemorrhage (Eye disorders) | 8 | 6
Vision Blurred (Eye disorders) | 10 | 2
Diarrhoea (Gastrointestinal disorders) | 70 | 103
Nausea (Gastrointestinal disorders) | 75 | 83
Constipation (Gastrointestinal disorders) | 65 | 60
Vomiting (Gastrointestinal disorders) | 39 | 33
Abdominal Pain (Gastrointestinal disorders) | 33 | 30
Abdominal Distension (Gastrointestinal disorders) | 18 | 17
Haemorrhoids (Gastrointestinal disorders) | 18 | 12
Stomatitis (Gastrointestinal disorders) | 14 | 16
Mouth Haemorrhage (Gastrointestinal disorders) | 16 | 8
Dry Mouth (Gastrointestinal disorders) | 11 | 12
Dyspepsia (Gastrointestinal disorders) | 14 | 9
Dysphagia (Gastrointestinal disorders) | 9 | 10
Gingival Bleeding (Gastrointestinal disorders) | 12 | 7
Oral Pain (Gastrointestinal disorders) | 5 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 9 | 4
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 9
Mouth Ulceration (Gastrointestinal disorders) | 9 | 2
Oedema Peripheral (General disorders) | 62 | 76
Fatigue (General disorders) | 53 | 53
Chills (General disorders) | 41 | 41
Mucosal Inflammation (General disorders) | 28 | 31
Pyrexia (General disorders) | 33 | 25
Asthenia (General disorders) | 14 | 14
Oedema (General disorders) | 13 | 14
Chest Pain (General disorders) | 11 | 13
Catheter Site Erythema (General disorders) | 9 | 7
Catheter Site Pain (General disorders) | 11 | 4
Chest Discomfort (General disorders) | 8 | 6
Pneumonia (Infections and infestations) | 28 | 26
Sepsis (Infections and infestations) | 5 | 8
Cellulitis (Infections and infestations) | 9 | 10
Bacteraemia (Infections and infestations) | 12 | 4
Transfusion Reaction (Injury, poisoning and procedural complications) | 13 | 14
Procedural Pain (Injury, poisoning and procedural complications) | 12 | 10
Fall (Injury, poisoning and procedural complications) | 12 | 8
Contusion (Injury, poisoning and procedural complications) | 9 | 11
Weight Decreased (Investigations) | 5 | 11
Decreased Appetite (Metabolism and nutrition disorders) | 50 | 62
Fluid Overload (Metabolism and nutrition disorders) | 13 | 19
Back Pain (Musculoskeletal and connective tissue disorders) | 22 | 21
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 20 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 9
Neck Pain (Musculoskeletal and connective tissue disorders) | 12 | 8
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 10 | 6
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 4 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Headache (Nervous system disorders) | 53 | 37
Dizziness (Nervous system disorders) | 32 | 31
Dysgeusia (Nervous system disorders) | 12 | 11
Somnolence (Nervous system disorders) | 3 | 9
Insomnia (Psychiatric disorders) | 36 | 38
Confusional State (Psychiatric disorders) | 20 | 26
Anxiety (Psychiatric disorders) | 23 | 22
Delirium (Psychiatric disorders) | 6 | 13
Depression (Psychiatric disorders) | 10 | 10
Hallucination (Psychiatric disorders) | 5 | 8
Agitation (Psychiatric disorders) | 8 | 4
Renal Failure Acute (Renal and urinary disorders) | 11 | 13
Haematuria (Renal and urinary disorders) | 10 | 10
Dysuria (Renal and urinary disorders) | 8 | 10
Pollakiuria (Renal and urinary disorders) | 8 | 8
Urinary Incontinence (Renal and urinary disorders) | 9 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 33
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 54 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36 | 32
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 30 | 30
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 26 | 29
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 28 | 16
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 12 | 14
Rales (Respiratory, thoracic and mediastinal disorders) | 12 | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Rash (Skin and subcutaneous tissue disorders) | 44 | 33
Petechiae (Skin and subcutaneous tissue disorders) | 21 | 18
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 13
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 14 | 13
Erythema (Skin and subcutaneous tissue disorders) | 14 | 10
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 | 13
Night Sweats (Skin and subcutaneous tissue disorders) | 14 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 17
Blood Blister (Skin and subcutaneous tissue disorders) | 14 | 5
Rash Pruritic (Skin and subcutaneous tissue disorders) | 10 | 6
Dry Skin (Skin and subcutaneous tissue disorders) | 8 | 7
Rash Erythematous (Skin and subcutaneous tissue disorders) | 6 | 8
Skin Lesion (Skin and subcutaneous tissue disorders) | 4 | 9
Hypotension (Vascular disorders) | 30 | 30
Hypertension (Vascular disorders) | 29 | 23
Deep Vein Thrombosis (Vascular disorders) | 8 | 9
Tachycardia (Cardiac disorders) | 22 | 17
Ecchymosis (Skin and subcutaneous tissue disorders) | 9 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No